CLINICAL TRIAL: NCT00153387
Title: Illinois WISEWOMAN Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-3949; 57-CCU520899-01
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: CVD Risk
MeSH Terms: interventions — Women's Health

INTERVENTIONS:
Behavioral: Women's health

SUMMARY:
To provide low-income, under- or uninsured 40- to 64-year-old women with the knowledge, skills, and opportunities to improve diet, physical activity, and other lifestyle behaviors to prevent, delay and control cardiovascular and other chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* NBCCEDP

Exclusion Criteria:

-

Ages: 40 Years to 64 Years | Sex: Female
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Julie Will, Study Chair — Centers for Disease Control and Prevention